CLINICAL TRIAL: NCT00766831
Title: Hydromorphone OROS in Korean Cancer Patients: Evaluation of Its Clinical Usefulness in Improvement of Sleep Disturbance
Brief Title: An Efficacy and Safety Study of Hydromorphone Oral Osmotic System (OROS) in Korean Participants With Cancer Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014806; HYD-KOR-4002
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-09

CONDITIONS: Cancer Pain
Keywords: Cancer pain; Hydromorphone OROS; Jurnista
MeSH Terms: conditions — Cancer Pain | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydromorphone OROS (Experimental): Participants will receive hydromorphone OROS (8 milligram [mg] up to greater than or equal to 32 mg) once daily for 2 weeks, in a dose adjusted according to previously administered strong oral opioid analgesic (dose with equivalent analgesic effect; hydromorphone OROS dose: oral morphine dose=1:5) hydromorphone OROS will be continued as per Investigator's discretion for additional 84 days of extension phase.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — Participants will receive hydromorphone OROS (8 milligram [mg] to greater than or equal to 32 mg) once daily for 2 weeks, in a dose adjusted according to previously administered strong oral opioid analgesic (dose with equivalent analgesic effect; hydromorphone OROS dose: oral morphine dose=1:5) hydromorphone OROS will be continued as per Investigator's discretion for additional 84 days of extension phase.
  Other Names: Jurnista

SUMMARY:
The purpose of this is study to evaluate improvement of sleep disorder caused by cancer pain after the administration of Hydromorphone Oral Osmotic System (OROS) in Korean participants with cancer.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (conducted in more than 1 center), prospective (study following participants forward in time) dose-ascending study to evaluate the clinical usefulness of hydromorphone OROS in improvement of sleep disturbance caused by cancer pain.Total duration of study will be 3 weeks. The study consists of 3 phases: Screening phase (up to 1 week), Treatment phase (2 weeks), and Extension phase (12 weeks). The study will include 6 visits: Day -7, Day 1, Day 15, Day 43, Day 71, and Day 99. During screening phase, potential participants will receive strong oral (long acting) opioid analgesic (for 7 days) until Day 1 and the participants will be evaluated for participation in clinical study on Day 1. During treatment phase, participants will receive hydromorphone OROS (8 milligram [mg] to greater than or equal to 32 mg), once daily for 2 weeks, and the dose will be adjusted every 2 days from Day 3 at the Investigator's discretion and according to the strong oral (long acting) opioid analgesic administered from screening phase to Day 1 (the initial dose of the study drug will be determined by converting the dose of the previously administered analgesic to that of the daily dose of oral morphine with the equivalent analgesic effect to the study drug [dose with equivalent analgesic effect; Hydromorphone OROS dose: oral morphine dose =1:5]). Participants who completed treatment phase and suffer from continuing cancer pain will be enrolled to extension phase and study drug will be administered as per Investigator discretion for 99 days. Participants primarily will be evaluated for improvement in sleep disturbance measured by Korean Brief Pain Inventory (KBPI). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are currently receiving strong opioid analgesic (drug used to control pain) for their cancer pain management
* Participants whose arithmetical mean of sleep disturbance caused by pain measured with Numeric Rating Scale for 3 days before Visit 2 (Day 1) is equal to or greater than 4 points
* Participants who are able, in the opinion of Investigator, to comply fully with the trial requirements including completion of the Korean-Brief Pain Inventory
* Participants who have signed an informed consent form

Exclusion Criteria:

* Participants with pain who are not likely to response to opioid analgesics
* Participants who are intolerant or hypersensitive to hydromorphone
* Participants with the following digestive tract diseases which is serious enough to interfere action of an oral analgesic; diseases which can affect absorption and transit of oral drugs such as dysphagia (trouble swallowing), vomiting, no bowel movement, intestinal obstruction, serious intestinal stenosis (narrowing of a duct, tube, or 1 of the valves in the heart), etc
* Female participants of childbearing potential who are pregnant or lactating, seeking pregnancy, or failing to take adequate contraceptive precautions
* Participants in whom the risks of treatment with morphine/hydromorphone outweigh the potential benefits, including such risk categories as raised intracranial pressure, hypotension, hypothyroidism, asthma, compromised respiratory function compromised liver function, convulsive (an involuntary contraction or series of contractions of the voluntary muscles) disorder and Addison disease (disorder that occurs when the adrenal glands do not produce enough of their hormones)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydromorphone OROS: Participants received hydromorphone oral osmotic system OROS (8 milligram [mg] to greater than or equal to 32 mg) once daily for 2 weeks, in a dose adjusted according to previously administered strong oral opioid analgesic (dose with equivalent analgesic effect; hydromorphone OROS dose: oral morphine dose=1:5) hydromorphone OROS was continued as per Investigator's discretion for additional 84 days of extension phase.
Period: Overall Study
Arm/Group | Hydromorphone OROS
Started | 190
Completed | 75
Not Completed | 115
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 20
Not completed — Protocol Violation | 15
Not completed — Physician Decision | 5
Not completed — Withdrawal of consent | 26
Not completed — Non cooperation by participants | 14
Not completed — Other | 28

BASELINE CHARACTERISTICS:
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 190
Age Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 129

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment Response in Sleep Disturbance Caused by Cancer Pain
Description: Percentage of treatment response in sleep disturbance caused by cancer pain was reported. Treatment response in sleep disturbance was measured by Numeric Rating Scale (NRS) ranging from 0=no disturbance to 10=extreme disturbance.
Time Frame: Day 15 or Early withdrawal
Population: Intent to treat (ITT) population included all the participants who received study medication at least 1 dose of study medication and had the data on sleep disturbance caused by pain at Day 15. Last observation carried forward (LOCF) was used.
Measure: Number (95% Confidence Interval); unit: Percentage of treatment response
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Percentage of treatment response | 34.9 [27.8 to 41.9]

2. Secondary Outcome: Sleep Disturbance Questionnaire: Analgesic Administration
Description: The Investigator evaluated sleep disturbance through the participant's answers to below question in "yes" or "no" response: 'Did you need to take an analgesic for pain relief in order to go to sleep last night?'
Time Frame: Baseline and Day 15
Population: ITT population included all the participants who received at least 1 dose of study medication and had the data on sleep disturbance caused by pain at Day 15. LOCF was used.
Measure: Number; unit: Participants
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Participants
  Baseline : Yes | 37
  Baseline: No | 45
  Day 15: Yes | 25
  Day 15: No | 57

3. Secondary Outcome: Sleep Disturbance Questionnaire: Frequency of Waking Up
Description: The Investigator evaluated sleep disturbance through the participant's answers to below question: How many times did you wake up while sleeping late night (frequency [once, 2 times, 3 times, 4 times, 5 times, couldn't fall asleep at all] of waking up due to pain last night).
Time Frame: Baseline and Day 15
Population: ITT population included all the participants who received at least 1 dose of study medication and had the data on sleep disturbance caused by pain at Day 15. LOCF was used. Here 'n' signifies participants who were evaluated for this outcome measure at a particular time point.
Measure: Number; unit: Participants
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Participants
  Baseline: once (n=77) | 8
  Baseline: 2 times (n=77) | 29
  Baseline: 3 times (n=77) | 21
  Baseline: 4 times (n=77) | 6
  Baseline: 5 times (n=77) | 13
  Day 15: once (n=58) | 23
  Day 15: 2 times (n=58) | 17
  Day 15: 3 times (n=58) | 7
  Day 15: 4 times (n=58) | 7
  Day 15: 5 times (n=58) | 4

4. Secondary Outcome: Sleep Disturbance Questionnaire: Wake up Due to Unbearable Pain
Description: The Investigator evaluated sleep disturbance through the participant's answers to below question in "yes" or "no" response: 'Did you wake up because of unbearable pain this morning?'
Time Frame: Baseline and Day 15
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Participants
  Baseline: Yes | 32
  Baseline: No | 50
  Day 15: Yes | 15
  Day 15: No | 67

5. Secondary Outcome: Korean Brief Pain Inventory (K-BPI) Questionnaire Score
Description: K-BPI is a questionnaire designed to measure the degree of pain severity and the impact of pain in performing daily routines. K-BPI comprises of 9 items out of which 6 items were assessed. Score of each item ranges from 0 to 10, where 0=no pain/impact and 10=severe pain/impact. The 6 items that were assessed are: a) level of pain worst in last 24 hours; b) level of pain weakest in last 24 hours; c) level of pain average in last 24 hours; d) level of pain right now; e) how much pain reduced with the therapy taken; sixth item was further classified into 7 categories: i) general activities ii) mood iii) ambulatory ability iv) routine works v) interpersonal relation vi) sleep vii) life enjoyment.
Time Frame: Baseline and Day 15
Population: ITT population included all the participants who received at least 1 dose of study medication and had the data on sleep disturbance caused by pain at Day 15. LOCF was used. Here 'n' signifies the number of participant who were evaluated for particular category at particular time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Units on a scale
  Baseline: Worst pain in last 24 hours (n=74) | 6.7 (1.9)
  Baseline: Weakest pain in last 24 hours (n=74) | 3.6 (2.1)
  Baseline: Average pain in last 24 hours (n=74) | 5.2 (1.6)
  Baseline: Level of pain right now (n=76) | 4.4 (1.8)
  Baseline: Pain reduced from therapy taken (n=76) | 0.4 (0.3)
  Baseline: General activities (n=76) | 5.0 (2.0)
  Baseline: Mood (n=76) | 5.1 (2.0)
  Baseline: Ambulatory ability (n=75) | 5.0 (2.3)
  Baseline: Routine works (n=76) | 5.6 (2.2)
  Baseline: Interpersonal relation (n=76) | 4.8 (2.6)
  Baseline: Sleep (n=76) | 5.9 (1.8)
  Baseline: Life enjoyment (n=76) | 5.5 (2.5)
  Day 15: Worst pain in last 24 hours (n=75) | 5.4 (2.0)
  Day 15: Weakest pain in last 24 hours (n=75) | 2.9 (1.9)
  Day 15: Average pain in last 24 hours (n=74) | 4.1 (1.9)
  Day 15: Level of pain right now (n=75) | 3.7 (2.0)
  Day 15: Pain reduced from therapy taken (n=75) | 0.5 (0.3)
  Day 15: General activities (n=75) | 5.0 (2.0)
  Day 15: Mood (n=75) | 4.6 (2.3)
  Day 15: Ambulatory ability (n=75) | 4.5 (2.6)
  Day 15: Routine works (n=75) | 4.9 (2.4)
  Day 15: Interpersonal relation (n=76) | 4.6 (2.7)
  Day 15: Sleep (n=74) | 4.2 (2.5)
  Day 15: Life enjoyment (n=75) | 5.0 (2.6)

6. Secondary Outcome: Participant's Pain Intensity
Description: Participant's pain intensity was measured using NRS ranging from 0=no pain to 10=unimaginable extreme pain. Participants maintained pain diary for 3 days before Baseline until Day 15 and pain intensity was measured twice daily (morning and afternoon). Here average pain intensity is reported. Average pain intensity was calculated as mean of morning pain intensity and evening pain intensity for each baseline and Day 15.
Time Frame: Baseline and Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Units on a scale
  Baseline | 5.3 (1.7)
  Day 15 | 4.1 (1.8)

7. Secondary Outcome: Number of Times the Short-Acting Opioid Analgesic Administered for Breakthrough Pain
Description: The participants recorded the frequency of short acting opioid analgesic taken for treating breakthrough pain among the pains suffered by the participants. Here frequency means number of times the short-acting opioid analgesic administered for breakthrough pain from baseline to Day 15
Time Frame: Baseline and Day 15
Population: ITT population included all the participants who received at least 1 dose of study medication and had the data on sleep disturbance caused by pain at Day 15. LOCF was used. Here 'N' signifies participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Frequency of breakthrough pain drug
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 76
Frequency of breakthrough pain drug
  Baseline | 0.92 (1.29)
  Day 15 | 0.36 (0.93)

8. Secondary Outcome: Number of Participants With Each Grade of Eastern Cooperative Oncology Group (ECOG) Performance Status Score
Description: The ECOG performance status was used to evaluate participant's disease progression and the effect of the disease on the participant's activities of daily living. ECOG performance status score ranges from Grade 0 to 4, where Grade 0=Fully active, Grade 1=restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, Grade 2=ambulatory and capable of all self-care but unable to carry out any work activities, Grade 3=capable of only limited self-care, confined to bed or chair, and Grade 4=completely disabled.
Time Frame: Baseline and Day 15
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Participants
  Baseline: Grade 0 | 1
  Baseline: Grade 1 | 53
  Baseline: Grade 2 | 23
  Baseline: Grade 3 | 4
  Baseline: Grade 4 | 1
  Day 15: Grade 1 | 52
  Day 15: Grade 2 | 22
  Day 15: Grade 3 | 5
  Day 15: Grade 4 | 3

9. Secondary Outcome: Number of Participants With Clinical Global Impression-Improvement (CGI-Improvement) Score
Description: The CGI-Improvement score evaluates how much the participant's condition is improved compared to Baseline. The score ranges from 1 to 7, where 1=improved very much, 2=Improved much, 3=Improved a little, 4=No change, 5=Aggravated a little,6=Aggravated much and 7=aggravated very much.
Time Frame: Day 15
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Participants
  Improved very much | 1
  Improved much | 21
  Improved a little | 37
  No change | 20
  Aggravated a little | 2
  Aggravated much | 1

10. Secondary Outcome: Number of Participants in Each Category of Global Assessment of Overall Efficacy of Study Drug Assessed by Participants
Description: Participants evaluated overall efficacy of study drug according to the rating of 1=not effective, 2=average, 3=effective, 4=very effective and 5=extremely effective.
Time Frame: Day 15
Population: ITT population included all the participants who received at least one dose of study medication and had the data on sleep disturbance caused by pain at Day 15. LOCF was used.
Measure: Number; unit: Participants
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Participants
  Not effective | 7
  Average | 29
  Effective | 38
  Very effective | 8

11. Secondary Outcome: Number of Participants in Each Category of Global Assessment of Overall Efficacy of Study Drug Assessed by Investigators
Description: Investigator evaluated overall efficacy of study drug according to the rating of 1=not effective, 2=average, 3=effective, 4=very effective and 5=extremely effective.
Time Frame: Day 15
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Participants
  Not effective | 7
  Average | 32
  Effective | 32
  Very effective | 10
  Extremely effective | 1

12. Secondary Outcome: Percentage of Participants Who Preferred the Oral Long-Action Opioids Analgesic or Study Drug
Description: Participant's preferences between the oral long-action opioids analgesic and the study drug was reported.
Time Frame: Day 15
Population: ITT population included all the participants who received at least one dose of study medicaation and had the data on sleep disturbance caused by pain at Day 15. Last observation carried forward (LOCF) was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Percentage of participants
  Hydromorphone hydrochloride OROS tablets | 80.5
  Previously administered strong opioid analgesic | 19.5

13. Secondary Outcome: Percentage of Participants With Different Reasons for Their Preference for Oral Long-Action Opioids Analgesic or Study Drug
Description: Participants reasons for preference between the long acting oral opioid analgesic and the study drug administered were reported. Reasonos for preferences were "I experienced a certain pain relief effect during the administration of the drug", "I didn't wake up due to pain while sleeping", "It was more convenient because the number of administrations was reduced", "I could reduce the administration of short acting narcotic analgesic to treat breakthrough pain" and "other".
Time Frame: Day 15
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Hydromorphone OROS
Number analyzed (Participants) | 82
Percentage of participants
  Hydromorphone OROS: pain relief | 1.5
  Previously administered analgesic: pain relief | 37.5
  Hydromorphone OROS: couldn't wake up | 31.8
  Previously administered analgesic:couldn | 50.0
  Hydromorphone OROS: reduced doses | 54.6
  Previously administered analgesic: reduced doses | 12.5
  Hydromorphone OROS: could reduce administration | 12.1
  Previously taken analgesic: reduce administration | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 15
Description: Safety analysis population included all the participants who received at least 1 dose of study medication
Arm/Group | Hydromorphone OROS
Serious Adverse Events (participants affected / at risk) | 22/120
Other Adverse Events (participants affected / at risk) | 90/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydromorphone OROS (N=120)
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
ileus (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 2
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Somnolence (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Disease progression (General disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hydromorphone OROS (N=120)
Constipation (Gastrointestinal disorders) | 50
Nausea (Gastrointestinal disorders) | 33
Vomiting (Gastrointestinal disorders) | 24
Diarrhoea (Gastrointestinal disorders) | 7
Somnolence (Nervous system disorders) | 61
Dizziness (Nervous system disorders) | 43
Asthenia (General disorders) | 45
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22
Pruritus (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No